CLINICAL TRIAL: NCT07144111
Title: A Phase 1, Open-Label, Single-Dose Study to Evaluate the Effect of Moderate or Severe Hepatic Impairment on the Pharmacokinetics of Inavolisib
Brief Title: A Study to Evaluate the Effect of Moderate or Severe Hepatic Impairment on the Pharmacokinetics (PK) of Inavolisib
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Genentech, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: GP45942
Record Dates: First submitted 2025-08-20; First posted 2025-08-27 (Actual); Last update posted 2026-02-12 (Actual); Status verified 2026-02

CONDITIONS: Hepatic Impairment
MeSH Terms: interventions — inavolisib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Cohort 1 (Experimental): Participants with normal hepatic function will receive a single oral dose of inavolisib on Day 1
  Interventions: Drug: Inavolisib
- Cohort 2 (Experimental): Participants with moderate hepatic function will receive a single oral dose of inavolisib on Day 1
  Interventions: Drug: Inavolisib
- Cohort 3 (Experimental): Participants with severe hepatic function will receive a single oral dose of inavolisib on Day 1
  Interventions: Drug: Inavolisib

INTERVENTIONS:
Drug: Inavolisib — Participants will receive a single oral dose of inavolisib

SUMMARY:
This open-label study will evaluate the effect on the pharmacokinetics (PK), safety, and tolerability of a single oral dose of inavolisib in participants with moderate or severe hepatic impairment compared with demographically matched healthy participants with normal hepatic function.

ELIGIBILITY:
Inclusion Criteria:

All participants:

* Body Mass Index 18.0 to 40.0 kilogram per meter square (kg/m^2), inclusive, and body weight >=45 kg.
* Negative hepatitis B surface antigen (HBsAg) test
* Positive hepatitis B surface antibody (HBsAb) test or negative HBsAb
* Negative HIV (Human Immunodeficiency Virus) test
* Females will not be pregnant or breastfeeding and must be either postmenopausal or surgically sterile
* Males will agree to use contraception and will refrain from sperm donation

Healthy participants (Cohort 1):

* Negative hepatitis C virus (HCV) antibody test or positive HCV antibody test followed by a negative HCV RNA test
* Normal hepatic function and no history of clinically significant hepatic dysfunction

Participants with Hepatic Impairment (Cohorts 2 and 3):

* Considered to have moderate (Child-Pugh score of 7 to 9) or severe (Child-Pugh score of 10 to 15) hepatic impairment
* Chronic, stable hepatic insufficiency with features of cirrhosis
* Negative hepatitis C viral load

Exclusion Criteria:

All participants:

* History of Type 1 diabetes or Type 2 Diabetes that is insulin-dependent or requires ongoing systemic treatment with two or more agents
* Significant history or clinical manifestation of any metabolic, allergic, dermatological, renal, hematological, pulmonary, cardiovascular, gastrointestinal (GI), neurological, or psychiatric disorder
* Significant illness, surgery, or hospitalization within 2 weeks prior to dosing.
* History of gastro-intestinal surgery
* Malabsorption syndrome or any other condition that would interfere with enteral absorption.
* History of active or latent Mycobacterium tuberculosis (TB), regardless of treatment history, or positive QuantiFERON® TB Gold test
* History of significant hypersensitivity, intolerance, or allergy to any drug compound, food, or other substance
* Use of drugs of abuse (including opioids)

Healthy participants (Cohort 1):

- History of alcoholism or drug addiction

Participants with Hepatic Impairment (Cohorts 2 and 3):

* Hepatic impairment due to hepatocellular carcinoma or bile duct cancer
* Surgical or artificial portosystemic shunt (e.g., transjugular intrahepatic portosystemic shunt)
* Evidence of hepatorenal syndrome
* Ascites requiring paracentesis
* Any evidence of progressive liver disease in the last 1 month
* Receipt of a liver transplant
* Hepatic encephalopathy Grade 2 or above

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 32 (Estimated)
Dates: Start 2025-08-21 (Actual); Primary Completion 2026-09-05 (Estimated); Study Completion 2026-09-09 (Estimated)

PRIMARY OUTCOMES:
Maximum Observed Concentration (Cmax) of Inavolisib | Pre-dose (0 hour), 30 minutes (min), 1, 1.5, 2, 3, 4, 6, 8, 10, 24, 48, 72, and 96 hours postdose
Area Under Curve (AUC) from Hour 0 to the Last Measurable Concentration (AUC [0-t]) of Inavolisib | Pre-dose (0 hour), 30 minutes (min), 1, 1.5, 2, 3, 4, 6, 8, 10, 24, 48, 72, and 96 hours postdose
AUC from Zero to Infinity (AUC [0-inf]) Extrapolated of Inavolisib | Pre-dose (0 hour), 30 minutes (min), 1, 1.5, 2, 3, 4, 6, 8, 10, 24, 48, 72, and 96 hours postdose
Geometric Mean Ratio of Cmax of Inavolisib | Pre-dose (0 hour), 30 minutes (min), 1, 1.5, 2, 3, 4, 6, 8, 10, 24, 48, 72, and 96 hours postdose
Geometric Mean Ratio of AUC (0-t) of Inavolisib | Pre-dose (0 hour), 30 minutes (min), 1, 1.5, 2, 3, 4, 6, 8, 10, 24, 48, 72, and 96 hours postdose
Geometric Mean Ratio of AUC (0-inf) of Inavolisib | Pre-dose (0 hour), 30 minutes (min), 1, 1.5, 2, 3, 4, 6, 8, 10, 24, 48, 72, and 96 hours postdose

SECONDARY OUTCOMES:
Percentage of Participants with Treatment Emergent Adverse Events (TEAEs) | From Baseline up to Follow-up (Day 8)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Genentech, Inc.
Locations (4):
- United States (4):
  - Orange County Research Center, Lake Forest, California
  - Orlando Clinical Research Center, Orlando, Florida
  - The Texas Liver Institute, Inc., San Antonio, Texas
  - Pinnacle Clinical Research - San Antonio, San Antonio, Texas

IPD SHARING:
Plan to Share IPD: No